CLINICAL TRIAL: NCT02571140
Title: A Phase Ib Study to Assess the Safety, Pharmacokinetics and Pharmacodynamics of Oral PTH (1-34) Formulations in Healthy Subjects
Brief Title: A Study to Assess the Safety, Pharmacokinetics and Pharmacodynamics of Oral PTH (1-34) Formulations in Healthy Subjects
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Entera Bio Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: ENT-02-2013
Record Dates: First submitted 2015-10-06; First posted 2015-10-08 (Estimated); Last update posted 2018-01-10 (Actual); Status verified 2018-01

CONDITIONS: Drug Safety and Bioavailability
MeSH Terms: interventions — Teriparatide; Parathyroid Hormone

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Active Comparator (Active Comparator): Subcutaneous injection of Teriparatide
  Interventions: Drug: Teriparatide
- Oral PTH (1-34) (Experimental): Oral administration of pill with API with different optimizations
  Interventions: Drug: Oral PTH (1-34)

INTERVENTIONS:
Drug: Teriparatide — subcutaneous standard injection
  Arms: Active Comparator
Drug: Oral PTH (1-34) — Different optimization of API
  Other Names: Teriparatide
  Arms: Oral PTH (1-34)

SUMMARY:
This study will have one stage consisting of multiple treatment visits. The study is designed to assess the safety and bioavailability of Entera's oral PTH(1 - 34) in adult male healthy volunteers in various formulation. The study is also designed to assess the reproducibility of pharmacokinetic profiles with various formulations.

ELIGIBILITY:
Inclusion Criteria:

1. Signed Informed consent to the study.
2. Males ,aged 18 - 50 years, BMI 18-30 kg/m2, inclusive,
3. Subjects able to adhere to the visit schedule and protocol requirements
4. Hematology ,Chemistry and Urinalysis values with no clinical significance or do not reflect a medical condition which according to the physicians' judgment might confound the results of the study or pose additional risk to the subject by participation in the study.
5. Hemoglobin level > 12.5 g/dl
6. Blood pressure levels with no clinical significance.
7. Negative serology to HIV, Hepatitis B, Hepatitis C.
8. No known drug and alcohol abuse
9. Negative urinary drugs of abuse at screening
10. No sensitivity to dairy products
11. No allergy to soy bean products.
12. No prescription medications taken within one month to enrollment
13. Over-the-counter drugs (including vitamins) taken within 14 days prior to visit 2 are subject to the investigators' discretion for inclusion.
14. No subjects with previous urolithiasis.
15. Non-smoking In good health as determined by past medical history, physical examination, vital signs, electrocardiogram and laboratory tests at screening

Exclusion Criteria:

1. Concurrent therapy that, in the Investigator's opinion, would interfere with the evaluation of the safety or efficacy of the study medication.
2. Treatment with any investigational product within the last 30 days, enrollment or intention to enroll in any active study involving the use of investigational devices or drugs.
3. Presence of any other condition or circumstance that, in the judgment of the Investigator, might increase the risk to the patient or decrease the chance of obtaining satisfactory data to achieve the objectives of the study.
4. Active infections
5. History of drug or alcohol abuse
6. Known allergies or sensitivities to components of study treatment or study procedures, including Soy.
7. Clinically diagnosed psychiatric disorders that may interfere with patient study participation
8. Medical history known or suspected to increase risks of AEs related to study drug, up to the investigator's discretion
9. Chronic illnesses, up to the investigator's discretion

Ages: 18 Years to 50 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 30 (Actual)
Dates: Start 2013-10; Primary Completion 2017-08 (Actual); Study Completion 2017-10 (Actual)

PRIMARY OUTCOMES:
Peak Plasma Concentration | 60-522 days
  Blood samples for determination of PTH plasma concentrations will be taken at the time points to study the pharmocokinetc profile

SECONDARY OUTCOMES:
Adverse Events | 60-522 days
  throughout the study beginning from the time the subject signs the consent form until the end of study, subjects will complete the following evaluations:
  Vital signs (blood pressure, heart rate, oral temperature) Clinical laboratory evaluations, hematology, chemistry Physical Exam ECG

CONTACTS AND LOCATIONS:
Overall Officials: Yosef Caraco, MD, Principal Investigator — Hadassah Ein Kerem Medical Center